CLINICAL TRIAL: NCT01263496
Title: A Long-term, Open-label Extension Study to Investigate the Long-term Safety of SYR-322 in Subjects With Type 2 Diabetes in Japan.
Brief Title: Long-term Safety Study of Alogliptin in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322/OCT-001; U1111-1118-4027 (Registry Identifier: WHO)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; voglibose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Alogliptin 6.25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 50 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Voglibose 0.2-mg TID (Active Comparator)
  Interventions: Drug: Voglibose

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 6.25 mg, tablets, orally, once daily for up to 40 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 6.25 mg QD
Drug: Alogliptin — Alogliptin 12.5 mg, tablets, orally, once daily for up to 40 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily for up to 40 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Alogliptin — Alogliptin 50 mg, tablets, orally, once daily for up to 40 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 50 mg QD
Drug: Voglibose — Voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  Other Names: Voglib; BASEN®
  Arms: Voglibose 0.2-mg TID

SUMMARY:
The purpose of this study was to evaluate the long-term safety and efficacy of SYR-322, once daily (QD), to an α-glucosidase inhibitor, three times daily (TID), administered for 40 consecutive weeks in participants who completed a phase 2 dose-ranging study.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

To evaluate the long-term safety and efficacy of alogliptin, this extension study was administered for 40 consecutive weeks (52 weeks from the start of treatment in the phase 2 dose-ranging study) to participants who had completed the phase 2 dose-ranging study SYR-322/CCT-001 (NCT01263470).

ELIGIBILITY:
Inclusion Criteria:

* Had completed the phase 2 dose-ranging study (i.e., the subject had completed the study visit at Week 12).

Exclusion Criteria:

* Had clinical manifestations of hepatic impairment (e.g., an aspartate aminotransferase or alanine aminotransferase value 2.5 times or more of the upper reference limit at Week 8 of treatment in the phase 2 dose-ranging study).
* Had clinical manifestations of renal impairment (e.g., a creatinine value of 2 mg/dL or more at Week 8 of treatment in the phase 2 dose-ranging study).

Ages: 29 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Department of Medicine, Study Director — Kawasaki Medical School

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 53 investigative sites in Japan from 10 May 2007 to 27 September 2008.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with uncontrolled blood glucose despite diet and exercise therapies were enrolled in one of 5, once-daily (QD) or three-times daily (TID) treatment groups.
  Analyses were performed by treatment dose group or by treatment dose in this study.
Groups:
- Alogliptin 6.25 mg Dose Group* → Alogliptin 6.25 mg Dose Group: Alogliptin 6.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the 6.5 mg dosing ARM of the SYR-322/CCT-001 (NCT01263470) dose-ranging study.
- Alogliptin 12.5 mg Dose Group* → Alogliptin 12.5 mg Dose Group: Alogliptin 12.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the 12.5 mg dosing ARM of the SYR-322/CCT-001 (NCT01263470) dose-ranging study.
- Alogliptin 25 mg Dose Group* → Alogliptin 25 mg Dose Group: Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the 25 mg dosing ARM of the SYR-322/CCT-001 (NCT01263470) dose-ranging study.
- Alogliptin 50 mg Dose Group* → Alogliptin 50 mg Dose Group: Alogliptin 50 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the 50 mg dosing ARM of the SYR-322/CCT-001 (NCT01263470) dose-ranging study.
- Voglibose 0.2 mg Dose Group* → Voglibose 0.2 mg Dose Group: Voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the voglibose 0.2 mg dosing ARM of the SYR-322/CCT-001 (NCT01263470) dose-ranging study.
- Placebo Dose Group* → Alogliptin 6.25 mg Dose Group; Placebo Dose Group* → Alogliptin 12.5 mg Dose Group; Placebo Dose Group* → Alogliptin 25 mg Dose Group; Placebo Dose Group* → Alogliptin 50 mg Dose Group: Placebo-matching tablets, orally, once or three times daily for up to 40 weeks.
  *for participants from the placebo dosing ARM of the SYR-322/CCT-001 (NCT01263470) dose-ranging study.
Period: Enrolled - Long-Term Extension Study
Arm/Group | Alogliptin 6.25 mg Dose Group* → Alogliptin 6.25 mg Dose Group | Alogliptin 12.5 mg Dose Group* → Alogliptin 12.5 mg Dose Group | Alogliptin 25 mg Dose Group* → Alogliptin 25 mg Dose Group | Alogliptin 50 mg Dose Group* → Alogliptin 50 mg Dose Group | Voglibose 0.2 mg Dose Group* → Voglibose 0.2 mg Dose Group | Placebo Dose Group* → Alogliptin 6.25 mg Dose Group | Placebo Dose Group* → Alogliptin 12.5 mg Dose Group | Placebo Dose Group* → Alogliptin 25 mg Dose Group | Placebo Dose Group* → Alogliptin 50 mg Dose Group
Started | 72 | 75 | 72 | 75 | 74 | 17 | 17 | 18 | 18
Completed | 71 | 75 | 72 | 74 | 72 | 17 | 17 | 18 | 18
Not Completed | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Period: Entered - Long-Term Extension Study
Arm/Group | Alogliptin 6.25 mg Dose Group* → Alogliptin 6.25 mg Dose Group | Alogliptin 12.5 mg Dose Group* → Alogliptin 12.5 mg Dose Group | Alogliptin 25 mg Dose Group* → Alogliptin 25 mg Dose Group | Alogliptin 50 mg Dose Group* → Alogliptin 50 mg Dose Group | Voglibose 0.2 mg Dose Group* → Voglibose 0.2 mg Dose Group | Placebo Dose Group* → Alogliptin 6.25 mg Dose Group | Placebo Dose Group* → Alogliptin 12.5 mg Dose Group | Placebo Dose Group* → Alogliptin 25 mg Dose Group | Placebo Dose Group* → Alogliptin 50 mg Dose Group
Started | 71 | 72 (3 participants did not enter from previous period (1 voluntary withdraw; 2 did not meet criteria).) | 72 | 74 | 71 (1 participant did not enter from previous period (voluntary withdraw).) | 17 | 17 | 17 (1 participant did not enter from previous period (voluntary withdraw).) | 18
Completed | 62 | 59 | 62 | 68 | 61 | 16 | 16 | 16 | 15
Not Completed | 9 | 13 | 10 | 6 | 10 | 1 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 5 | 6 | 3 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 2 | 4 | 1 | 1 | 0 | 1
Not completed — Lack of Efficacy | 8 | 4 | 4 | 1 | 5 | 0 | 0 | 0 | 1
Not completed — Participant Unavailability | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alogliptin 6.25 mg QD: Alogliptin 6.25 mg, tablets, orally, once daily for up to 40 weeks.
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily for up to 40 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily for up to 40 weeks.
- Alogliptin 50 mg QD: Alogliptin 50 mg, tablets, orally, once daily for up to 40 weeks.
- Voglibose 0.2 mg TID: Voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID | Total
Number analyzed (Participants) | 96 | 101 | 97 | 97 | 83 | 474
Age, Customized [Number; unit: participants]
  ≤ 64 years | 69 | 67 | 64 | 65 | 51 | 316
  ≥ 65 years | 27 | 34 | 33 | 32 | 32 | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 22 | 29 | 27 | 133
  Male | 70 | 72 | 75 | 68 | 56 | 341

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pre-treatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug, which increases in intensity after the start of dosing. Adverse events data with onset occurring more than 30 days after last dose of study drug (AE start date - last dose date >30) will be listed, but not included in the summary tables below.
Time Frame: 52 Weeks.
Population: Adverse Event Profile in the Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 96 | 101 | 97 | 97 | 83
participants
  Serious Adverse Event | 1 | 5 | 8 | 5 | 4
  Serious Adverse Event Related to Study Drug | 1 | 2 | 2 | 2 | 0
  Other Adverse Events (Incidence ≥3%) | 78 | 81 | 81 | 88 | 74

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 94 | 94 | 79
percentage of Glycosylated Hemoglobin | -0.55 (0.703) | -0.70 (0.545) | -0.74 (0.520) | -0.86 (0.499) | -0.15 (0.735)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.401, 95% CI 2-sided [-0.618 to -0.184]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.548, 95% CI 2-sided [-0.739 to -0.358]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.590, 95% CI 2-sided [-0.779 to -0.401]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.708, 95% CI 2-sided [-0.894 to -0.522]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 88 | 89 | 89 | 91 | 71
percentage of Glycosylated Hemoglobin | -0.57 (0.758) | -0.75 (0.586) | -0.77 (0.616) | -0.90 (0.565) | -0.25 (0.633)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.316, 95% CI 2-sided [-0.538 to -0.093]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.493, 95% CI 2-sided [-0.684 to -0.302]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.510, 95% CI 2-sided [-0.706 to -0.314]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.647, 95% CI 2-sided [-0.834 to -0.461]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 87 | 87 | 88 | 90 | 69
percentage of Glycosylated Hemoglobin | -0.56 (0.699) | -0.69 (0.628) | -0.70 (0.672) | -0.88 (0.602) | -0.30 (0.650)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.263, 95% CI 2-sided [-0.479 to -0.047]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.395, 95% CI 2-sided [-0.598 to -0.192]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.405, 95% CI 2-sided [-0.616 to -0.195]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.583, 95% CI 2-sided [-0.780 to -0.386]

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 24).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 86 | 84 | 89 | 89 | 66
percentage of Glycosylated Hemoglobin | -0.47 (0.736) | -0.61 (0.697) | -0.66 (0.714) | -0.83 (0.647) | -0.29 (0.730)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.172, 95% CI 2-sided [-0.410 to 0.065]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.319, 95% CI 2-sided [-0.550 to -0.088]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.370, 95% CI 2-sided [-0.601 to -0.139]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.533, 95% CI 2-sided [-0.752 to -0.314]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 28).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 28 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 85 | 82 | 87 | 86 | 65
percentage of Glycosylated Hemoglobin | -0.39 (0.804) | -0.56 (0.721) | -0.67 (0.749) | -0.78 (0.705) | -0.32 (0.676)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.079, 95% CI 2-sided [-0.323 to 0.166]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.241, 95% CI 2-sided [-0.471 to -0.011]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.357, 95% CI 2-sided [-0.590 to -0.124]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.467, 95% CI 2-sided [-0.692 to -0.242]

7. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 32).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 32 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 84 | 81 | 87 | 85 | 64
percentage of Glycosylated Hemoglobin | -0.35 (0.787) | -0.56 (0.811) | -0.61 (0.777) | -0.76 (0.757) | -0.27 (0.662)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.080, 95% CI 2-sided [-0.321 to 0.162]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.294, 95% CI 2-sided [-0.542 to -0.046]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.341, 95% CI 2-sided [-0.579 to -0.103]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.487, 95% CI 2-sided [-0.722 to -0.252]

8. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 36).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 36 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 82 | 81 | 82 | 84 | 64
percentage of Glycosylated Hemoglobin | -0.33 (0.724) | -0.52 (0.857) | -0.66 (0.722) | -0.77 (0.759) | -0.28 (0.664)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.279 to 0.182]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.234, 95% CI 2-sided [-0.491 to 0.023]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.375, 95% CI 2-sided [-0.605 to -0.145]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.488, 95% CI 2-sided [-0.724 to -0.252]

9. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 40).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 40 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 81 | 79 | 79 | 84 | 63
percentage of Glycosylated Hemoglobin | -0.33 (0.686) | -0.48 (0.882) | -0.66 (0.694) | -0.77 (0.765) | -0.28 (0.627)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.050, 95% CI 2-sided [-0.270 to 0.169]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.193, 95% CI 2-sided [-0.453 to 0.067]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.374, 95% CI 2-sided [-0.596 to -0.152]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.490, 95% CI 2-sided [-0.723 to -0.256]

10. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 44).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 44 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 65 | 61 | 63 | 69 | 63
percentage of Glycosylated Hemoglobin | -0.29 (0.649) | -0.59 (0.722) | -0.71 (0.767) | -0.79 (0.770) | -0.35 (0.632)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.065, 95% CI 2-sided [-0.160 to 0.289]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.236, 95% CI 2-sided [-0.477 to 0.005]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.360, 95% CI 2-sided [-0.608 to -0.113]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.435, 95% CI 2-sided [-0.679 to -0.191]

11. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 48).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 48 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 63 | 60 | 62 | 69 | 61
percentage of Glycosylated Hemoglobin | -0.43 (0.590) | -0.66 (0.716) | -0.76 (0.736) | -0.83 (0.779) | -0.40 (0.695)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Net) = -0.033, 95% CI 2-sided [-0.262 to 0.196]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.262, 95% CI 2-sided [-0.516 to -0.008]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.358, 95% CI 2-sided [-0.614 to -0.103]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.432, 95% CI 2-sided [-0.690 to -0.174]

12. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 52).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 62 | 59 | 62 | 68 | 61
percentage of Glycosylated Hemoglobin | -0.49 (0.544) | -0.65 (0.726) | -0.74 (0.754) | -0.85 (0.785) | -0.37 (0.723)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.118, 95% CI 2-sided [-0.346 to 0.110]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.277, 95% CI 2-sided [-0.539 to -0.015]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.373, 95% CI 2-sided [-0.637 to -0.109]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.477, 95% CI 2-sided [-0.741 to -0.213]

13. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Final Visit).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 96 | 101 | 96 | 97 | 83
percentage of Glycosylated Hemoglobin | -0.40 (0.713) | -0.47 (0.817) | -0.63 (0.788) | -0.86 (0.723) | -0.22 (0.882)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.181, 95% CI 2-sided [-0.416 to 0.055]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.245, 95% CI 2-sided [-0.492 to 0.003]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.408, 95% CI 2-sided [-0.654 to -0.161]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.638, 95% CI 2-sided [-0.874 to -0.402]

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 94 | 94 | 79
mg/dL | -12.1 (32.26) | -15.3 (23.57) | -17.0 (21.42) | -23.0 (23.35) | -3.6 (26.98)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.51, 95% CI 2-sided [-17.56 to 0.54]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -11.70, 95% CI 2-sided [-19.23 to -4.18]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -13.41, 95% CI 2-sided [-20.68 to -6.15]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -19.38, 95% CI 2-sided [-26.93 to -11.83]

15. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 16).
Description: The change between the value of fasting plasma glucose collected at week 16 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 88 | 89 | 89 | 97 | 71
mg/dL | -10.8 (24.52) | -15.8 (23.76) | -17.0 (23.34) | -18.8 (29.74) | -6.4 (28.02)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -4.44, 95% CI 2-sided [-12.67 to 3.80]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -9.39, 95% CI 2-sided [-17.48 to -1.30]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -10.56, 95% CI 2-sided [-18.58 to -2.54]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -12.37, 95% CI 2-sided [-21.44 to -3.31]

16. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 20).
Description: The change between the value of fasting plasma glucose collected at week 20 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 87 | 87 | 88 | 90 | 69
mg/dL | -11.5 (27.50) | -15.3 (24.49) | -13.8 (23.10) | -20.1 (27.94) | -4.6 (27.53)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.90, 95% CI 2-sided [-15.66 to 1.86]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -10.73, 95% CI 2-sided [-18.97 to -2.49]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -9.21, 95% CI 2-sided [-17.20 to -1.23]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -15.49, 95% CI 2-sided [-24.27 to -6.72]

17. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 24).
Description: The change between the value of fasting plasma glucose collected at week 24 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 86 | 84 | 89 | 89 | 66
mg/dL | -10.6 (29.15) | -11.7 (28.19) | -13.8 (23.70) | -20.2 (28.90) | -8.3 (25.58)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.27, 95% CI 2-sided [-11.22 to 6.67]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-12.16 to 5.44]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.43, 95% CI 2-sided [-13.30 to 2.44]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -11.90, 95% CI 2-sided [-20.74 to -3.06]

18. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 28).
Description: The change between the value of fasting plasma glucose collected at week 28 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 85 | 82 | 87 | 86 | 65
mg/dL | -9.6 (30.07) | -13.4 (30.06) | -14.1 (23.86) | -19.9 (32.36) | -7.2 (28.13)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.44, 95% CI 2-sided [-11.97 to 7.08]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.25, 95% CI 2-sided [-15.84 to 3.35]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.93, 95% CI 2-sided [-15.28 to 1.41]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -12.73, 95% CI 2-sided [-22.67 to -2.78]

19. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 32).
Description: The change between the value of fasting plasma glucose collected at week 32 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 84 | 81 | 87 | 85 | 64
mg/dL | -14.5 (21.13) | -12.9 (31.64) | -14.9 (25.86) | -20.3 (30.72) | -9.1 (26.59)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.44, 95% CI 2-sided [-13.19 to 2.31]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.77, 95% CI 2-sided [-13.53 to 5.99]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.85, 95% CI 2-sided [-14.36 to 2.67]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -11.22, 95% CI 2-sided [-20.72 to -1.73]

20. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 36).
Description: The change between the value of fasting plasma glucose collected at week 36 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 81 | 82 | 81 | 84 | 64
mg/dL | -10.7 (24.25) | -14.3 (32.31) | -16.9 (23.66) | -20.9 (32.48) | -8.4 (25.36)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.26, 95% CI 2-sided [-10.42 to 5.90]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.90, 95% CI 2-sided [-15.64 to 3.84]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.47, 95% CI 2-sided [-16.52 to -0.42]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -12.47, 95% CI 2-sided [-22.18 to -2.76]

21. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 40).
Description: The change between the value of fasting plasma glucose collected at week 40 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 81 | 79 | 79 | 84 | 63
mg/dL | -13.5 (19.32) | -14.8 (28.76) | -15.7 (21.38) | -23.2 (29.40) | -13.8 (25.82)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-7.10 to 7.77]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-10.16 to 8.21]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-9.71 to 5.95]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -9.38, 95% CI 2-sided [-18.59 to -0.18]

22. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 44).
Description: The change between the value of fasting plasma glucose collected at week 44 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 65 | 61 | 63 | 69 | 63
mg/dL | -16.7 (22.28) | -18.7 (26.79) | -19.0 (24.77) | -24.7 (29.69) | -15.0 (26.09)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-10.20 to 6.75]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-13.10 to 5.70]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.97, 95% CI 2-sided [-12.94 to 5.00]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -9.74, 95% CI 2-sided [-19.40 to -0.08]

23. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 48).
Description: The change between the value of fasting plasma glucose collected at week 48 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 62 | 60 | 62 | 69 | 61
mg/dL | -16.0 (21.54) | -20.8 (24.97) | -22.8 (21.89) | -25.4 (30.50) | -13.5 (26.30)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-11.00 to 6.15]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -7.29, 95% CI 2-sided [-16.53 to 1.94]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -9.30, 95% CI 2-sided [-17.93 to -0.67]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -11.88, 95% CI 2-sided [-21.83 to -1.93]

24. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 52).
Description: The change between the value of fasting plasma glucose collected at week 52 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 62 | 59 | 62 | 68 | 61
mg/dL | -13.7 (21.54) | -19.5 (25.63) | -21.4 (22.35) | -26.0 (29.05) | -12.5 (25.77)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-9.68 to 7.27]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -7.05, 95% CI 2-sided [-16.34 to 2.24]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.86, 95% CI 2-sided [-17.47 to -0.26]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -13.51, 95% CI 2-sided [-23.12 to -3.89]

25. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Final Visit).
Description: The change between the value of fasting plasma glucose collected at week 52 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 96 | 101 | 96 | 97 | 83
mg/dL | -10.4 (27.13) | -15.5 (31.02) | -17.1 (26.50) | -27.6 (28.13) | -8.8 (30.14)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-10.09 to 6.80]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -6.70, 95% CI 2-sided [-15.66 to 2.25]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.28, 95% CI 2-sided [-16.64 to 0.07]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -18.82, 95% CI 2-sided [-27.39 to -10.24]

26. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 12).
Description: The change between the value of fasting C-peptide collected at week 12 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 94 | 94 | 79
ng/mL | -0.02 (0.667) | 0.19 (0.604) | 0.19 (0.567) | 0.25 (0.706) | -0.04 (0.900)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.219 to 0.254]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.226, 95% CI 2-sided [0.002 to 0.451]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.230, 95% CI 2-sided [0.008 to 0.453]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.282, 95% CI 2-sided [0.041 to 0.524]

27. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 16).
Description: The change between the value of fasting C-peptide collected at week 16 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 88 | 89 | 89 | 91 | 71
ng/mL | 0.08 (0.790) | 0.22 (0.640) | 0.33 (0.679) | 0.46 (0.924) | -0.01 (0.886)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.173 to 0.353]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.228, 95% CI 2-sided [-0.010 to 0.467]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.339, 95% CI 2-sided [0.095 to 0.584]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.468, 95% CI 2-sided [0.184 to 0.752]

28. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 20).
Description: The change between the value of fasting C-peptide collected at week 20 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 86 | 86 | 88 | 90 | 69
ng/mL | 0.15 (0.634) | 0.35 (0.781) | 0.28 (0.608) | 0.56 (0.971) | -0.16 (0.953)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.317, 95% CI 2-sided [0.064 to 0.570]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.511, 95% CI 2-sided [0.236 to 0.786]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.437, 95% CI 2-sided [0.190 to 0.685]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.718, 95% CI 2-sided [0.413 to 1.022]

29. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 24).
Description: The change between the value of fasting C-peptide collected at week 24 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 83 | 80 | 83 | 85 | 66
ng/mL | 0.12 (0.742) | 0.26 (0.722) | 0.20 (0.603) | 0.23 (0.620) | -0.10 (0.831)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.226, 95% CI 2-sided [-0.029 to 0.481]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.358, 95% CI 2-sided [0.104 to 0.612]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.308, 95% CI 2-sided [0.076 to 0.540]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.331, 95% CI 2-sided [0.098 to 0.565]

30. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 28).
Description: The change between the value of fasting C-peptide collected at week 28 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 80 | 73 | 77 | 80 | 65
ng/mL | 0.11 (0.692) | 0.21 (0.642) | 0.26 (0.591) | 0.29 (0.857) | -0.04 (0.951)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [-0.130 to 0.410]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.245, 95% CI 2-sided [-0.026 to 0.516]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.294, 95% CI 2-sided [0.035 to 0.552]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.329, 95% CI 2-sided [0.032 to 0.626]

31. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 32).
Description: The change between the value of fasting C-peptide collected at week 32 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 67 | 66 | 74 | 73 | 63
ng/mL | 0.03 (0.778) | 0.41 (0.652) | 0.45 (0.718) | 0.37 (0.816) | -0.01 (0.950)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [-0.252 to 0.349]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.420, 95% CI 2-sided [0.138 to 0.703]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.460, 95% CI 2-sided [0.178 to 0.742]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.384, 95% CI 2-sided [0.085 to 0.683]

32. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 36).
Description: The change between the value of fasting C-peptide collected at week 36 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 55 | 46 | 50 | 54 | 48
ng/mL | 0.12 (0.714) | 0.33 (0.639) | 0.20 (0.750) | 0.42 (0.856) | 0.09 (0.777)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.257 to 0.326]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.249, 95% CI 2-sided [-0.043 to 0.542]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [-0.196 to 0.417]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.333, 95% CI 2-sided [0.010 to 0.656]

33. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 40).
Description: The change between the value of fasting C-peptide collected at week 40 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 33 | 26 | 35 | 41 | 35
ng/mL | -0.14 (0.998) | 0.48 (0.836) | 0.27 (0.735) | 0.44 (0.567) | 0.13 (1.066)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.268, 95% CI 2-sided [-0.769 to 0.233]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.349, 95% CI 2-sided [-0.156 to 0.855]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [-0.297 to 0.577]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.308, 95% CI 2-sided [-0.075 to 0.690]

34. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 44).
Description: The change between the value of fasting C-peptide collected at week 44 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 17 | 18 | 20 | 20 | 21
ng/mL | 0.22 (0.963) | 0.52 (0.887) | 0.59 (0.881) | 0.20 (0.651) | -0.06 (0.991)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.281, 95% CI 2-sided [-0.367 to 0.928]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.579, 95% CI 2-sided [-0.035 to 1.194]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.647, 95% CI 2-sided [0.054 to 1.241]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.252, 95% CI 2-sided [-0.280 to 0.785]

35. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 48).
Description: The change between the value of fasting C-peptide collected at week 48 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 6 | 7 | 9 | 6 | 9
ng/mL | -0.40 (0.632) | 0.54 (0.796) | 0.04 (0.485) | 0.15 (0.558) | -0.10 (0.934)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.300, 95% CI 2-sided [-1.246 to 0.646]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.643, 95% CI 2-sided [-0.305 to 1.591]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [-0.599 to 0.888]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.250, 95% CI 2-sided [-0.673 to 1.173]

36. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 52).
Description: The change between the value of fasting C-peptide collected at week 52 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 2 | 3 | 3 | 4 | 3
ng/mL | -0.25 (0.212) | 0.73 (0.874) | 0.10 (0.781) | 0.30 (1.095) | 0.70 (1.473)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.950, 95% CI 2-sided [-4.462 to 2.562]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-2.712 to 2.779]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.600, 95% CI 2-sided [-3.273 to 2.073]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.400, 95% CI 2-sided [-2.874 to 2.074]

37. Secondary Outcome: Change From Baseline in Fasting C-peptide (Final Visit).
Description: The change between the value of fasting C-peptide collected at week 52 or final visit and fasting C-peptide collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 96 | 101 | 96 | 97 | 83
ng/mL | 0.34 (1.046) | 0.44 (0.820) | 0.32 (0.805) | 0.48 (0.765) | 0.18 (0.970)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [-0.140 to 0.458]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.260, 95% CI 2-sided [-0.001 to 0.520]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.136, 95% CI 2-sided [-0.126 to 0.398]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.298, 95% CI 2-sided [0.042 to 0.553]

38. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Week 12).
Description: The change between the value of blood glucose collected at week 12 and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 95 | 94 | 79
mg/dL | 62.9 (33.75) | 61.8 (31.41) | 56.4 (36.70) | 55.8 (30.83) | 64.8 (31.62)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-11.82 to 7.99]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.02, 95% CI 2-sided [-12.45 to 6.40]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.41, 95% CI 2-sided [-18.77 to 1.96]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -8.96, 95% CI 2-sided [-18.35 to 0.44]

39. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Week 24).
Description: The change between the value of blood glucose collected at week 24 and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 71 | 68 | 74 | 74 | 67
mg/dL | 64.3 (37.80) | 55.5 (30.63) | 55.5 (39.78) | 55.9 (33.60) | 56.6 (30.02)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 7.66, 95% CI 2-sided [-3.88 to 19.19]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-11.41 to 9.24]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-12.91 to 10.75]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-11.32 to 9.99]

40. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Week 52).
Description: The change between the value of blood glucose collected at week 52 and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 80 | 76 | 78 | 83 | 61
mg/dL | 65.7 (38.39) | 62.6 (30.18) | 58.3 (32.62) | 51.8 (36.73) | 61.0 (30.16)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 4.70, 95% CI 2-sided [-7.09 to 16.49]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [-8.63 to 11.89]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-13.36 to 7.98]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -9.20, 95% CI 2-sided [-20.58 to 2.17]

41. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Final Visit).
Description: The change between the value of blood glucose collected at week 52 or final visit and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 95 | 94 | 79
mg/dL | 65.0 (37.48) | 63.8 (32.46) | 60.4 (35.09) | 52.6 (37.07) | 52.6 (32.38)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-11.44 to 9.84]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-11.74 to 7.66]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.44, 95% CI 2-sided [-15.62 to 4.75]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -13.28, 95% CI 2-sided [-23.83 to -2.74]

42. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Week 12).
Description: as for outcome 38
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg·hr/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 95 | 94 | 79
mg·hr/dL | -57.0 (75.68) | -55.4 (61.17) | -67.8 (55.52) | -80.5 (51.95) | -50.0 (62.49)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -7.02, 95% CI 2-sided [-28.15 to 14.10]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -5.45, 95% CI 2-sided [-23.93 to 13.02]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -17.80, 95% CI 2-sided [-35.46 to -0.13]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -30.58, 95% CI 2-sided [-47.75 to -13.41]

43. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Week 24).
Description: as for outcome 39
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg·hr/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 70 | 68 | 74 | 74 | 67
mg·hr/dL | -43.9 (76.23) | -52.5 (74.32) | -69.8 (73.23) | -75.1 (68.57) | -62.4 (62.68)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 18.45, 95% CI 2-sided [-5.18 to 42.09]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 9.86, 95% CI 2-sided [-13.56 to 33.28]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -7.44, 95% CI 2-sided [-30.25 to 15.37]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -12.80, 95% CI 2-sided [-34.75 to 9.15]

44. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Week 52).
Description: as for outcome 40
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg·hr/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 80 | 76 | 78 | 83 | 61
mg·hr/dL | -59.5 (50.66) | -62.0 (59.52) | -69.0 (64.88) | -88.7 (73.36) | -65.4 (67.93)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 5.84, 95% CI 2-sided [-13.90 to 25.58]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 3.35, 95% CI 2-sided [-18.20 to 24.90]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -3.64, 95% CI 2-sided [-26.03 to 18.74]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -23.37, 95% CI 2-sided [-47.08 to 0.34]

45. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Final Visit).
Description: as for outcome 41
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg·hr/dL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 95 | 94 | 79
mg·hr/dL | -53.5 (70.32) | -55.1 (76.72) | -67.6 (69.49) | -91.3 (71.93) | -56.4 (73.88)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 2.97, 95% CI 2-sided [-18.77 to 24.71]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [-21.21 to 23.94]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -11.20, 95% CI 2-sided [-32.69 to 10.30]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -34.90, 95% CI 2-sided [-56.85 to -12.96]

46. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Week 12).
Description: The change between the value of C-peptide collected at week 12 and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 97 | 95 | 94 | 79
ng·hr/mL | 0.56 (1.765) | 0.97 (1.975) | 0.96 (2.073) | 0.99 (1.742) | -0.39 (2.091)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.955, 95% CI 2-sided [0.375 to 1.535]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.358, 95% CI 2-sided [0.752 to 1.965]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.350, 95% CI 2-sided [0.724 to 1.975]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.380, 95% CI 2-sided [0.804 to 1.955]

47. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Week 24).
Description: The change between the value of C-peptide collected at week 24 and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 69 | 68 | 72 | 74 | 67
ng·hr/mL | 0.93 (2.068) | 1.35 (1.928) | 1.14 (1.743) | 1.38 (1.934) | -0.10 (1.994)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.034, 95% CI 2-sided [0.344 to 1.723]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.448, 95% CI 2-sided [0.780 to 2.115]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.243, 95% CI 2-sided [0.616 to 1.870]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.481, 95% CI 2-sided [0.827 to 2.136]

48. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Week 52).
Description: The change between the value of C-peptide collected at week 52 and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 6 | 4 | 3 | 5 | 3
ng·hr/mL | 1.91 (2.922) | 3.44 (3.320) | 2.37 (5.399) | 3.14 (2.368) | 1.86 (0.293)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [-4.088 to 4.188]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.585, 95% CI 2-sided [-3.476 to 6.647]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.517, 95% CI 2-sided [-8.151 to 9.184]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.277, 95% CI 2-sided [-2.191 to 4.744]

49. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Final Visit).
Description: The change between the value of C-peptide collected at week 52 or final visit and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 92 | 97 | 95 | 94 | 79
ng·hr/mL | 0.99 (2.087) | 1.45 (2.257) | 1.14 (2.054) | 1.41 (2.028) | 0.15 (1.866)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.841, 95% CI 2-sided [0.239 to 1.443]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.304, 95% CI 2-sided [0.679 to 1.930]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.992, 95% CI 2-sided [0.400 to 1.585]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.263, 95% CI 2-sided [0.674 to 1.853]

50. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Week 12).
Description: The change between the value of insulin collected at week 12 and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 86 | 94 | 85 | 90 | 68
μU·hr/mL | 0.49 (18.988) | 2.63 (15.416) | 4.44 (13.637) | -0.03 (21.572) | -15.40 (20.416)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 15.891, 95% CI 2-sided [9.597 to 22.184]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 18.026, 95% CI 2-sided [12.466 to 23.585]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 19.838, 95% CI 2-sided [14.379 to 25.297]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 15.368, 95% CI 2-sided [8.677 to 22.060]

51. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Week 24).
Description: The change between the value of insulin collected at week 24 and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 61 | 64 | 68 | 71 | 59
μU·hr/mL | -1.89 (21.943) | 4.50 (12.876) | 2.85 (12.309) | -0.98 (27.457) | -16.21 (20.927)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 14.323, 95% CI 2-sided [6.567 to 22.079]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 20.714, 95% CI 2-sided [14.563 to 26.864]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 19.063, 95% CI 2-sided [13.125 to 25.002]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 15.233, 95% CI 2-sided [6.618 to 23.847]

52. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Week 52).
Description: The change between the value of insulin collected at week 52 and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 76 | 70 | 75 | 80 | 56
μU·hr/mL | -7.62 (19.526) | -1.71 (15.032) | -0.44 (14.871) | -2.30 (22.985) | -15.66 (20.026)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 8.047, 95% CI 2-sided [1.169 to 14.924]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 13.950, 95% CI 2-sided [7.767 to 20.133]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 15.221, 95% CI 2-sided [9.191 to 21.251]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 13.366, 95% CI 2-sided [5.847 to 20.885]

53. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Final Visit).
Description: The change between the value of insulin collected at week 52 or final visit and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 87 | 91 | 91 | 91 | 70
μU·hr/mL | -6.93 (18.945) | -1.67 (15.508) | 0.43 (14.532) | -1.56 (21.843) | -14.65 (19.322)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 7.719, 95% CI 2-sided [1.657 to 13.782]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 12.978, 95% CI 2-sided [7.556 to 18.399]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 15.076, 95% CI 2-sided [9.808 to 20.345]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 13.087, 95% CI 2-sided [6.561 to 19.614]

54. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Week 12).
Description: The change between the value of glucagons collected at week 12 and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 92 | 96 | 95 | 93 | 79
pg·hr/mL | -9.5 (38.86) | -4.4 (36.89) | -6.6 (46.85) | -15.5 (41.23) | -16.3 (52.26)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 6.76, 95% CI 2-sided [-7.03 to 20.55]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 11.85, 95% CI 2-sided [-1.49 to 25.19]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 9.72, 95% CI 2-sided [-5.12 to 24.56]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-13.26 to 14.90]

55. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Week 24).
Description: The change between the value of glucagons collected at week 24 and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 70 | 67 | 74 | 74 | 67
pg·hr/mL | -1.7 (37.90) | 3.0 (41.66) | 0.9 (50.56) | -0.8 (43.71) | -7.6 (60.64)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 5.90, 95% CI 2-sided [-11.11 to 22.91]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 10.57, 95% CI 2-sided [-7.21 to 28.35]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 8.45, 95% CI 2-sided [-10.08 to 26.98]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 6.82, 95% CI 2-sided [-10.67 to 24.30]

56. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Week 52).
Description: The change between the value of glucagons collected at week 52 and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 80 | 75 | 78 | 82 | 61
pg·hr/mL | -10.7 (47.21) | -11.3 (45.41) | -14.5 (59.39) | -12.5 (52.10) | -13.8 (61.15)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 3.09, 95% CI 2-sided [-14.95 to 21.13]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [-15.61 to 20.57]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-21.00 to 19.68]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-17.47 to 20.05]

57. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Final Visit).
Description: The change between the value of glucagons collected at week 52 or final visit and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 93 | 96 | 95 | 93 | 79
pg·hr/mL | -9.8 (45.93) | -9.0 (48.99) | -10.3 (61.18) | -14.6 (51.22) | -13.9 (58.84)
Statistical Analysis 1: Comparison: Alogliptin 6.25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 4.08, 95% CI 2-sided [-11.70 to 19.86]
Statistical Analysis 2: Comparison: Alogliptin 12.5 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 4.94, 95% CI 2-sided [-11.14 to 21.03]
Statistical Analysis 3: Comparison: Alogliptin 25 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 3.65, 95% CI 2-sided [-14.42 to 21.73]
Statistical Analysis 4: Comparison: Alogliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-17.24 to 15.89]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 6.25 mg QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Alogliptin 50 mg QD | Voglibose 0.2 mg TID
Serious Adverse Events (participants affected / at risk) | 2/96 | 8/101 | 8/97 | 5/97 | 4/83
Other Adverse Events (participants affected / at risk) | 78/96 | 81/101 | 81/97 | 88/97 | 74/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 6.25 mg QD (N=96) | Alogliptin 12.5 mg QD (N=101) | Alogliptin 25 mg QD (N=97) | Alogliptin 50 mg QD (N=97) | Voglibose 0.2 mg TID (N=83)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 6.25 mg QD (N=96) | Alogliptin 12.5 mg QD (N=101) | Alogliptin 25 mg QD (N=97) | Alogliptin 50 mg QD (N=97) | Voglibose 0.2 mg TID (N=83)
Nasopharyngitis (Infections and infestations) | 29 | 29 | 32 | 34 | 21
Bronchitis (Infections and infestations) | 4 | 6 | 1 | 4 | 1
Gastroenteritis (Infections and infestations) | 2 | 2 | 4 | 3 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 2 | 2 | 3
Tinea pedis (Infections and infestations) | 2 | 1 | 0 | 2 | 3
Cystitis (Infections and infestations) | 2 | 0 | 0 | 3 | 2
Rhinitis (Infections and infestations) | 2 | 0 | 3 | 2 | 0
Seasonal allergy (Immune system disorders) | 7 | 5 | 3 | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 1
Headache (Nervous system disorders) | 6 | 0 | 7 | 3 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 5 | 1
Hypoaesthesia (Nervous system disorders) | 5 | 1 | 1 | 1 | 4
Cerebral infarction (Nervous system disorders) | 0 | 0 | 3 | 1 | 0
Cataract (Eye disorders) | 5 | 2 | 2 | 2 | 2
Diabetic retinopathy (Eye disorders) | 3 | 2 | 1 | 2 | 1
Conjunctivitis allergic (Eye disorders) | 3 | 0 | 0 | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 3
Hypertension (Vascular disorders) | 0 | 2 | 3 | 1 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 7 | 7 | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 4 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 4 | 6 | 8
Dental caries (Gastrointestinal disorders) | 4 | 4 | 2 | 6 | 5
Flatulence (Gastrointestinal disorders) | 2 | 4 | 1 | 2 | 8
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 4 | 2 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3 | 5 | 2
Gastritis (Gastrointestinal disorders) | 2 | 3 | 1 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 4
Periodontal disease (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 5 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 4 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 6 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 4 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 4 | 3 | 8 | 6
Alanine aminotransferase increased (Investigations) | 0 | 4 | 3 | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 0 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 1 | 2 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.